CLINICAL TRIAL: NCT02257632
Title: A Randomized, Single-blinded, Multicenter, Phase IV Study to Compare Systemic VEGF Protein Dynamics Following Monthly Intravitreal Injections of 0.5 mg Ranibizumab Versus 2 mg Aflibercept Until Study Week 12 in Patients With Neovascular (Wet) Age-related Macular Degeneration
Brief Title: Systemic Vascular Endothelial Growth Factor (VEGF) Protein Dynamics Following Intravitreal Injections of Ranibizumab Versus Aflibercept in Patients With Neovascular Age-related Macular Degeneration
Acronym: TIDE AMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRFB002ADE27
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-01

CONDITIONS: Wet Age-Related Macular Degeneration
MeSH Terms: interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 6 monthly intravitreal injections of 0.5 mg ranibizumab
  Interventions: Drug: Ranibizumab 0.5 mg
- Group 2 (Experimental): 3 monthly intravitreal injections of 2 mg aflibercept followed by 3 monthly intravitreal injections of 0.5 mg ranibizumab
  Interventions: Drug: Ranibizumab 0.5 mg; Drug: Aflibercept 2 mg

INTERVENTIONS:
Drug: Ranibizumab 0.5 mg — Administered as an intravitreal injection
  Other Names: Lucentis
Drug: Aflibercept 2 mg — Administered as an intravitreal injection
  Other Names: Eylea
  Arms: Group 2

SUMMARY:
The purpose of the study was to compare the effect of intravitreal injections of ranibizumab and aflibercept on systemic VEGF protein levels in treatment naïve wet neovascular Age-related Macular Degeneration (wAMD) patients in a detailed time course.

DETAILED DESCRIPTION:
A planned study visit schedule was established at the time of baseline visit (day 1) for all patients. Study assessments for patients were performed at screening visit, baseline (day 1), day 2, day 8 (± 1 day to allow for flexibility in scheduling) and as of day 15 through to day 169 at biweekly visits.

ELIGIBILITY:
Inclusion Criteria:

* Visual impairment predominantly due to neovascular AMD.
* Active, newly diagnosed, untreated, angiographically documented, CNV lesion (i.e. leakage on fluorescein angiography plus intraretinal, subretinal or sub-RPE fluid on OCT) secondary to neovascular AMD in line with SmPC of ranibizumab and aflibercept

Exclusion Criteria:

* Stroke or myocardial infarction less than 3 months prior to screening.
* Presence of uncontrolled systolic blood pressure or diastolic blood pressure
* Type 1 or Type 2 diabetes mellitus
* Use of any systemic anti-VEGF drugs
* Use of systemic or inhaled corticosteroids for at least 30 consecutive days within 3 months prior to screening.
* Women who are pregnant or breast feeding or who are menstruating and capable of becoming pregnant* and not practicing a medically approved method of contraception

For either eye:

* Any active periocular or ocular infection or inflammation
* Uncontrolled glaucoma
* Neovascularization of the iris or neovascular glaucoma
* History of treatment with any anti-angiogenic drugs

For study eye:

* Atrophy or fibrosis involving the center of the fovea at the time of screening or baseline.
* Cataract (if causing significant visual impairment), planned cataract surgery during the study period, vitrectomy, aphakia, glaucoma surgery, severe vitreous hemorrhage, rhegmatogenous retinal detachment, proliferative retinopathy or choroidal neovascularization of any other cause than wAMD
* Irreversible structural damage within 0.5 disc diameter of the center of the macula
* Any intraocular procedure (including cataract surgery, Yttrium-Aluminum-Garnet capsulotomy) within 3 months prior to baseline or anticipated within the next 6 months following baseline.
* Use of intravitreal or topical ocular corticosteroids administered for at least 30 consecutive days within 3 months prior to screening.

For fellow eye

- Retinal or choroidal neovascularization or macula edema of any cause

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Germany (5):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Regensburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included adult patients with active, newly diagnosed, and untreated wAMD. A total of 40 patients were treated at 6 study sites across Germany. Patients were treated in an outpatient setting.
Pre-assignment Details: At Screening, the eligibility criteria were performed.
  .
Groups:
- Ranibizumab: 6 monthly intravitreal injections of 0.5 mg ranibizumab
- Aflibercept and Ranibizumab: 3 monthly intravitreal injections of 2 mg aflibercept followed by 3 monthly intravitreal injections of 0.5 mg ranibizumab
Period: Overall Study
Arm/Group | Ranibizumab | Aflibercept and Ranibizumab
Started (All randomized patients) | 19 | 22
Full Analysis Set (FAS) (all randomized patients who received study treatment and had ≥ 1 primary efficacy assessment) | 19 | 21
Safety Set (SAF) (all patients who received study treatment and had ≥ 1 post-baseline safety assessment.) | 19 | 21
Per-Protocol Set (PPS) (all patients in the FAS who did not have any major protocol deviations) | 17 | 20
Completed | 18 | 19
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Aflibercept and Ranibizumab | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.3 (5.50) | 75.4 (8.94) | 74.9 (7.43)
Sex/Gender, Customized [Number; unit: Participants] — Population: Full Analysis Set (FAS)
  Participants
    Female | 11 | 10 | 21
    Male | 8 | 11 | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Standardized Area Under the Curve (AUC) for VEGF A Levels by SIMOA (Quanterix's Single Molecule Array) Method for the Comparative Phase
Description: The AUC was calculated using the trapezoidal rule, where all available measurement between Day 1 and Week 12 were used. The AUC was standardized by dividing the calculated value by the number of days from first to last measurement.
Time Frame: Baseline up to Week 12 visit (Days 1, 2, 8, 15, 29, 43, 57, 71, 85)
Population: Per-Protocol Set (PPS)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ranibizumab | Aflibercept and Ranibizumab
Number analyzed (Participants) | 17 | 20
pg/mL | 18.78 (8.460) | 33.95 (7.659)
Statistical Analysis 1: Comparison: Ranibizumab vs Aflibercept and Ranibizumab; Test type: Superiority; p < 0.0001, ANCOVA — missing Baseline VEGF-A level covariate values were imputed by the mean value of non-missing Baseline VEGF-A level from all other patients; including treatment group and center as fixed effect factors and Baseline VEGF-A as a covariate; Mean Difference (Final Values) = -14.98, 95% CI 2-sided [-19.64 to -10.32]

2. Secondary Outcome: Systemic VEGF-A Protein Levels From Study Week 12 to 24
Description: Systemic VEGF-A protein levels in patients switching from monthly 2 mg aflibercept injections to monthly 0.5 mg ranibizumab compared to patients treated with monthly 0.5 mg ranibizumab from baseline (standardized area under the curve)
Time Frame: From study week 12 to 24 (Days 85, 99, 113, 127, 141, 155, 169)
Population: Per-Protocol Set (PPS)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ranibizumab | Aflibercept and Ranibizumab
Number analyzed (Participants) | 17 | 20
pg/mL | 17.93 (5.316) | 29.07 (7.863)
Statistical Analysis 1: Comparison: Ranibizumab vs Aflibercept and Ranibizumab; Test type: Superiority; p < 0.0001, ANCOVA — missing Baseline VEGF-A level covariate values were imputed by the mean value of non-missing Baseline VEGF-A level from all the patients with values; including treatment group and center as fixed effect factors and Baseline VEGF-A as a covariate; Mean Difference (Final Values) = -11.46, 95% CI 2-sided [-15.98 to -6.94]

3. Secondary Outcome: Systemic VEGF-A Levels From Study Week 12 to 24 (Change From Baseline)
Description: Adjustment of systemic VEGF-A levels of patients switching from aflibercept to ranibizumab to levels comparable to baseline or to levels comparable as in patients treated from baseline with ranibizumab
Time Frame: From study week 12 to 24
Population: Per-Protocol Set (PPS) Number of participants analyzed at each time point represents patients with a value for both baseline and the specific post-baseline visit
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ranibizumab | Aflibercept and Ranibizumab
Number analyzed (Participants) | 17 | 20
pg/ml
  Change from Baseline at Week 12: number analyzed (Participants) | 16 | 17
  Change from Baseline at Week 12 | -1.37 (5.369) | 23.73 (13.700)
  Change from Baseline at Week 14: number analyzed (Participants) | 16 | 17
  Change from Baseline at Week 14 | -1.00 (6.128) | 21.93 (15.638)
  Change from Baseline at Week 16: number analyzed (Participants) | 15 | 15
  Change from Baseline at Week 16 | -0.01 (4.675) | 19.26 (16.432)
  Change from Baseline at Week 18: number analyzed (Participants) | 14 | 14
  Change from Baseline at Week 18 | 1.99 (5.582) | 11.61 (10.844)
  Change from Baseline at Week 20: number analyzed (Participants) | 15 | 16
  Change from Baseline at Week 20 | 1.62 (6.460) | 4.84 (11.065)
  Change from Baseline at Week 22: number analyzed (Participants) | 14 | 15
  Change from Baseline at Week 22 | 0.66 (8.109) | 2.45 (8.543)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 14
  Change from Baseline at Week 24 | -1.18 (3.664) | 0.96 (9.553)

ADVERSE EVENTS:
Time Frame: 28 weeks
Groups:
- Ranibizumab (Up to Month 3); Ranibizumab (After Month 3): 3 monthly intravitreal injections of 0.5 mg ranibizumab
- Aflibercept and Ranibizumab (Up to Month 3 - Aflibercept): 3 monthly intravitreal injections of 2 mg aflibercept (AEs reported that started before switching to ranibizumab)
- Aflibercept and Ranibizumab (After Month 3 - Ranibizumab): 3 monthly intravitreal injections of 0.5 mg ranibizumab (AEs reported that started on or after switching to ranibizumab)
Arm/Group | Ranibizumab (Up to Month 3) | Ranibizumab (After Month 3) | Aflibercept and Ranibizumab (Up to Month 3 - Aflibercept) | Aflibercept and Ranibizumab (After Month 3 - Ranibizumab)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/19 | 0/19 | 1/21 | 3/21
Other Adverse Events (participants affected / at risk) | 14/19 | 9/19 | 17/21 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (Up to Month 3) (N=19) | Ranibizumab (After Month 3) (N=19) | Aflibercept and Ranibizumab (Up to Month 3 - Aflibercept) (N=21) | Aflibercept and Ranibizumab (After Month 3 - Ranibizumab) (N=21)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Optic nerve cupping (Eye disorders) | 0 | 0 | 0 | 1
Retinal pigment epithelial tear (Eye disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (Up to Month 3) (N=19) | Ranibizumab (After Month 3) (N=19) | Aflibercept and Ranibizumab (Up to Month 3 - Aflibercept) (N=21) | Aflibercept and Ranibizumab (After Month 3 - Ranibizumab) (N=21)
Aortic valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 0 | 0
Anterior chamber cell (Eye disorders) | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0
Choroidal neovascularisation (Eye disorders) | 0 | 0 | 1 | 2
Conjunctival erosion (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 3 | 1 | 5 | 2
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 2 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 0
Macular fibrosis (Eye disorders) | 1 | 0 | 0 | 0
Metamorphopsia (Eye disorders) | 1 | 0 | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 1 | 0
Pinguecula (Eye disorders) | 1 | 0 | 0 | 0
Retinal fibrosis (Eye disorders) | 0 | 0 | 1 | 1
Retinal scar (Eye disorders) | 0 | 1 | 0 | 0
Subretinal fluid (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 2
Vitreous floaters (Eye disorders) | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fibrosis (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 1 | 0 | 1 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin E present (Investigations) | 1 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 1 | 2
Mean cell haemoglobin concentration increased (Investigations) | 1 | 0 | 0 | 0
Mean cell haemoglobin increased (Investigations) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Melanosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Jaw operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-04-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT02257632/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT02257632/SAP_001.pdf